CLINICAL TRIAL: NCT00093704
Title: EBV as Therapeutic Target: A Pilot Study of Inducing and Targeting EBV-TK in EBV-Positive Lymphomas by Combination of Bortezomib and Ganciclovir
Brief Title: Bortezomib and Ganciclovir in Treating Patients With Relapsed or Refractory Epstein Barr Virus-Positive Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: study could not recruit any more patients
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000389476; UCLA-0403021-01; MILLENNIUM-VEL-04-108; MILLENNIUM-EBV-NHL-01
Record Dates: First submitted 2004-10-06; First posted 2004-10-08 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2012-08

CONDITIONS: Lymphoma; Lymphoproliferative Disorder
Keywords: recurrent adult Hodgkin lymphoma; recurrent adult Burkitt lymphoma; post-transplant lymphoproliferative disorder; recurrent adult grade III lymphomatoid granulomatosis; angioimmunoblastic T-cell lymphoma; adult grade III lymphomatoid granulomatosis
MeSH Terms: conditions — Lymphoma; Lymphoproliferative Disorders; Hodgkin Disease; Burkitt Lymphoma; Immunoblastic Lymphadenopathy | interventions — Bortezomib; Ganciclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bortezomib + ganciclovir (Experimental): Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8 and 11. Patients also receive ganciclovir IV twice daily on days 1-14. Treatment repeats every 21 days for a maximum of 3 courses.
  Interventions: Drug: bortezomib + ganciclovir

INTERVENTIONS:
Drug: bortezomib + ganciclovir — Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8 and 11. Patients also receive ganciclovir IV twice daily on days 1-14. Treatment repeats every 21 days for a maximum of 3 courses.

SUMMARY:
RATIONALE: Bortezomib may stop the growth of cancer cells by blocking the enzymes necessary for their growth. The Epstein Barr virus can cause cancer and lymphoproliferative disorders. Ganciclovir is an antiviral drug that acts against the Epstein Barr virus. Giving ganciclovir together with bortezomib may kill more Epstein Barr virus-infected cancer cells.

PURPOSE: This clinical trial is studying how well giving bortezomib together with ganciclovir works in treating patients with relapsed or refractory Epstein Barr virus-positive lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Maximum Tolerated Dose (MTD) of bortezomib in patients with relapsed or refractory Epstein Barr virus-positive lymphoma.

Secondary

* Assess the antitumor effect of this regimen in these patients.

OUTLINE: This is a pilot, open-label, dose-escalation study of bortezomib.

Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8 and 11. Patients also receive ganciclovir IV twice daily on days 1-14. Treatment repeats every 21 days for a maximum of 3 courses.

Cohorts of 3-6 patients receive escalating doses of bortezomib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 3-9 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed Epstein Barr virus-positive lymphoma, including the following subtypes:

  * Post-transplantation lymphoma
  * Burkitt's lymphoma
  * Hodgkin's lymphoma
  * T-/NK-cell lymphoma
* Unresponsive to, or relapsed after, at least 1 prior chemotherapy regimen
* Bidimensionally measurable disease by CT scan
* At least 1 lesion ≥ 1.5 cm in the greatest diameter
* Age 18 and over
* ECOG 0-2 OR
* Karnofsky 50-100%
* Life expectancy More than 3 months
* Hematopoietic

  * Absolute neutrophil count ≥ 1,000/mm^3 (no growth factor support within the past 4 weeks)
  * Hemoglobin ≥ 9.0 g/dL
  * Platelet count ≥ 50,000/mm^3 (no platelet transfusions within the past 4 weeks)
* Hepatic

  * Bilirubin ≤ 2.0 times upper limit of normal (ULN)
  * AST and ALT ≤ 2.5 times ULN (5 times ULN in patients with liver involvement)
  * No active hepatitis B or C
* Renal

  * Creatinine clearance ≥ 60 mL/min
  * Sodium > 130 mmol/L
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* At least 4 weeks since prior immunotherapy
* At least 4 weeks since prior chemotherapy
* At least 4 weeks since prior radiotherapy
* More than 4 weeks since prior major surgery unless fully recovered
* Recovered from all prior therapy
* At least 4 weeks since prior investigational agents

Exclusion Criteria:

* primary or secondary CNS lymphoma or HIV-related lymphoma
* known brain metastases
* myocardial infarction within the past 6 months
* acute ischemia or new conduction system abnormalities by electrocardiogram
* symptomatic congestive heart failure
* unstable angina pectoris
* cardiac arrhythmia
* hospitalized
* pregnant or nursing
* other uncontrolled illness
* ongoing or active systemic infection
* psychiatric illness or social situation that would preclude study compliance
* history of allergic reaction attributable to compounds of similar chemical or biological composition to study drugs
* sensitivity to boron, mannitol, bortezomib, or ganciclovir
* concurrent corticosteroids (≥ 10 mg of prednisone or equivalent)
* concurrent radiotherapy
* other concurrent anticancer therapy
* other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2005-03; Primary Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
MTD of Bortezomib in patients with relapsed or refractory EBV + lymphomas | 3 weeks

SECONDARY OUTCOMES:
Bortezomib in inducing lytic gene expression in EBV-infected lymphoma cells | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sven De Vos, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States